CLINICAL TRIAL: NCT01872598
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Phase 3 Study to Evaluate the Safety and Efficacy of Masitinib in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Masitinib in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB09004
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; dementia; cognitive disease; memory loss; cerebrovascular disease; tyrosine kinase inhibitor
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognition Disorders; Memory Disorders; Cerebrovascular Disorders | interventions — masitinib; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Masitinib escalating dose (Experimental): Participants receive masitinib at 4.5 mg/kg/day, given orally twice daily, with a dose escalation to 6 mg/kg/day after 3 months of treatment
  Interventions: Drug: Masitinib; Drug: Standard of care
- Masitinib fixed dose (4.5 mg/kg/day) (Experimental): Participants receive masitinib at 4.5 mg/kg/day, given orally twice daily.
  Interventions: Drug: Masitinib; Drug: Standard of care
- Masitinib fixed dose (3.0 mg/kg/day) (Experimental): Participants receive masitinib at 3.0 mg/kg/day, given orally twice daily.
  Interventions: Drug: Masitinib; Drug: Standard of care
- Placebo (escalating dose) (Placebo Comparator): Participants receive placebo, given orally twice daily, with a matched dose escalation after 3 months of treatment
  Interventions: Drug: Placebo; Drug: Standard of care
- Placebo (fixed dose) (Placebo Comparator): Participants receive fixed dose placebo, given orally twice daily
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib escalating dose; Masitinib fixed dose (3.0 mg/kg/day); Masitinib fixed dose (4.5 mg/kg/day)
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo (escalating dose); Placebo (fixed dose)
Drug: Standard of care — stable dose of cholinesterase inhibitor (donepezil, rivastigmine or galantamine) and/or memantine, as per standard practice.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of masitinib for the treatment of mild to moderate Alzheimer's Disease. Masitinib will be administered as add-on therapy in patients who have been treated for a minimum of 6 months with a stable dose of cholinesterase inhibitor (donepezil, rivastigmine or galantamine) and/or memantine.

DETAILED DESCRIPTION:
Actual standard treatment for mild to moderately severe Alzheimer's dementia includes acetylcholinesterase inhibitors (donepezil, rivastigmine and galantamine) and a NMDA receptor antagonist (memantine for moderate to severe Alzheimer's disease). These medications have shown to have an effect on some cognitive and non cognitive symptoms of the pathology. However, their efficacy remains limited and may decrease with time. There is an unmet medical need in this pathology. Masitinib is a selective tyrosine kinase inhibitor that is thought to exert a neuroprotective effect through its activity on mast cells and other non-neuronal cells of the central nervous system, with subsequent modulation of inflammatory and neurodegenerative processes, as well as possibly disruption of the Aβ signaling cascade via inhibition of the Fyn signaling pathway. This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group study of oral masitinib. The objective of this study is to compare the efficacy and safety of masitinib at various doses versus matched placebo in the treatment of patients with mild to moderate Alzheimer's Disease. Masitinib will be administered as add-on therapy in patients who have been treated for a minimum of 6 months with a stable dose of cholinesterase inhibitor (donepezil, rivastigmine or galantamine) and/or memantine. Approximately 675 patients will be randomized into 5 treatment groups. The co-primary outcome measures are the Alzheimer's Disease Cooperative Study Activities of Daily Living score (ADCS-ADL), and Alzheimer's Disease Assessment Scale-Cognitive Subscale score (ADAS-Cog) after 24 weeks of treatment.

ELIGIBILITY:
Inclusion criteria include:

1. Patient with dementia of Alzheimer's type, according to the Diagnostic and Statistical Manual of Mental Disorders criteria (DSM-IV)
2. Patient with probable Alzheimer' disease according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association criteria (NINCDS-ADRDA)
3. Patient with MMSE ≥ 12 and ≤ 25 at baseline
4. Patient treated for a minimum of 6 months with a stable dose of cholinesterase inhibitors (donepezil, rivastigmine or galantamine) at baseline, and/or a stable dose of memantine for a minimum of 6 months at baseline, with no changes foreseen in therapy throughout the study.

Exclusion criteria include:

1. Patient with any other cause of dementia not due to Alzheimer's disease.
2. Patient with Alzheimer disease with severe forms of delusions or delirium (patients with light and mild forms of delusions and delirium will be allowed in the study).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
ADCS-ADL | 24 weeks
  Change in the Alzheimer's Disease Cooperative Study Activities of Daily Living score (ADCS-ADL).
ADAS-Cog | 24 weeks
  Change in the Alzheimer's Disease Assessment Scale-Cognitive Subscale score (ADAS-Cog).

SECONDARY OUTCOMES:
MMSE | 24 weeks
  Change in Mini Mental State Examination (MMSE)
CIBIC-plus | 24 weeks
  Clinician's Interview Based Impression of Change-plus (CIBIC-plus)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno DUBOIS, M.D., Ph.D., Principal Investigator — Pitié-Salpétrière
Locations (6):
- MHAT Sveta Marina, Varna, Bulgaria
- General Hospital of Thessaloniki, Thessaloniki, Greece
- Centrum Zdrowia Stołeczna 7, Bialystok, Poland
- Spitalul Universitar de Urgenta Elias, Bucharest, Romania
- Hospital Universitario Ramón y Cajal, Madrid, Spain
- Municipal Institution Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnikov, Dnipropetrovsk, Ukraine

REFERENCES:
- [Derived] Dubois B, Lopez-Arrieta J, Lipschitz S, Doskas T, Spiru L, Moroz S, Venger O, Vermersch P, Moussy A, Mansfield CD, Hermine O, Tsolaki M; AB09004 Study Group Investigators. Masitinib for mild-to-moderate Alzheimer's disease: results from a randomized, placebo-controlled, phase 3, clinical trial. Alzheimers Res Ther. 2023 Feb 28;15(1):39. doi: 10.1186/s13195-023-01169-x. PMID 36849969